CLINICAL TRIAL: NCT03807726
Title: Empower Breastfeeding: Effects of an Integrated Breastfeeding Education Program on Optimal Breastfeeding Practice
Brief Title: Empower Breastfeeding Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: N201701060
Record Dates: First submitted 2018-09-10; First posted 2019-01-17 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2018-04

CONDITIONS: Breastfeeding
Keywords: Breastfeeding, self-efficacy, education, intervention
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial with a two-arm design will be conducted among new mothers and their partners. The objectives are to determine whether an integrated breastfeeding education program based on breastfeeding self-efficacy theory [28, 31] will increase exclusive breastfeeding duration among women and psychological correlates of exclusive breastfeeding. This is a novel educational intervention incorporated simulation-based courses, mindfulness training, and professional support for targeting mother and her partner's self-efficacy enhancement.
Who Masked: Participant
Masking Description: Eligible participants will be randomly assigned to either intervention group or control group. A permuted block randomization method will be used to ensure equal number of subjects in each group. A block size of 4 including 6 different combinations, i.e., AABB, ABAB, ABBA, BBAA, BABA, and BAAB will be adopted. The sequence of block number will be generated randomly by the computer and then apply to the first four subjects and so on. The allocation concealment will be maintained by using opaque sealed envelopes containing the sequence number and will be prepared by the researcher who is not involved in participants' recruitment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Both standard usual care and the integrated breastfeeding education program (IBEP) will be provided to the participants in the intervention group. The integrated interventions are consisted of 1) four sessions of simulation breastfeeding education to build up the participants' performance accomplishment and vicarious learning including breastfeeding knowledge, skill, and self-efficacy; 2) two sessions of breastfeeding mindfulness training to equip women and their partners with stress reduction skills for their emotional arousal during breastfeeding; 3) a series of postpartum professional support to offer verbal persuasion in enhancing their breastfeeding skills and levels of self-efficacy. The details of each education components are presented at the following section.
  Interventions: Behavioral: Simulation breastfeeding education
- Control Group (No Intervention): The mother and her partner in the control group will receive the standard usual care provided at the study site. The study site hospital where follows the 10 steps of the Baby Friendly Hospital Initiative will provide breastfeeding care during prenatal check-up and postpartum care. The standard care protocols encompass elements such as prenatal breastfeeding consultation using breastfeeding pamphlets, and postpartum care like skin to skin contact, rooming- in, and breastfeeding consultation using pamphlets. The pregnant women need to register for childbirth class which contains only one breastfeeding class by themselves if needed. After delivery, the mothers are taught on breastfeeding knowledge and skills by the nurses at the postpartum ward or nursey.

INTERVENTIONS:
Behavioral: Simulation breastfeeding education — The integrated interventions are consisted of 1) four sessions of simulation breastfeeding education to build up the participants' performance accomplishment and vicarious learning including breastfeeding knowledge, skill, and self-efficacy; 2) two sessions of breastfeeding mindfulness training to equip women and their partners with stress reduction skills for their emotional arousal during breastfeeding; 3) a series of postpartum professional support to offer verbal persuasion in enhancing their breastfeeding skills and levels of self-efficacy.
  Other Names: Breastfeeding mindfulness training; Postpartum professional and partner support
  Arms: Intervention Group

SUMMARY:
This study results of integrated breastfeeding education program (IBEP) will guide in designing a theory-based breastfeeding educational module on promotion of optimal breastfeeding practice in new mother and her partner. The current novel education curriculum incorporated breastfeeding simulation, mindfulness training, and professional support will provide important information in supporting use of IBEP in enhancing participants self-efficacy. This study will show on how simulation teaching and mindfulness training can be utilized in the field of perinatal teaching to achieve better health outcomes.

DETAILED DESCRIPTION:
To achieve optimal breastfeeding practice, the development of an integrated breastfeeding education program (IBEP) which incorporates simulation education, mindfulness training, professional support targeting the self-efficacy of participants is of vital importance. A randomized controlled trial of an integrated breastfeeding education program focusing on participants will be designed with two study objectives: 1) to evaluate the effects of IBEP on the primary outcome measures of breastfeeding practice as following: a) early initiation of breastfeeding, b) exclusive breastfeeding rate, c) predominate breastfeeding rate; 2) to examine the effects of IBEP on the secondary outcome measures, psychosocial correlates of exclusive breastfeeding including a) breastfeeding self-efficacy, b)anxiety, c) depression, d) mindful awareness e) infant feeding attitude. These objectives will be examined among participants in six time periods: a) during pregnancy 24 to 32 weeks education program b) 34 to 40 weeks of pregnancy (after class or third trimester), c)1 week, d) 4weeks, d) 3 months, e) 6 months postpartum, while the indicators of breastfeeding practice will be examined at the four periods following delivery.

It is hypothesized that 1) the intervention will result in a better effect on all primary outcome measures, as compared to those in the control group. Specifically, participants in IBEP group will show 10 % or greater difference in exclusive breastfeeding rates at six months than participants in the control group, 2) participants in the IBEP group will demonstrate larger effects on breastfeeding self-efficacy and mindfulness, and lower anxiety and depression than those in the control group.

ELIGIBILITY:
Inclusion Criteria:

Aged 20 years and above. During the first or second trimester of pregnancy. Willing to breastfeed after delivery Singleton pregnancy. Participants are able to attend the breastfeeding class.

Exclusion Criteria:

Chronic medical conditions. Abnormal fetal screening. Preterm delivery before 37 weeks gestational weeks.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-18 (Actual); Study Completion 2019-05-18 (Actual)

PRIMARY OUTCOMES:
Breastfeeding self-efficacy | Change from Baseline Breastfeeding self-efficacy at 6 months.
  The Taiwanese version of the Breastfeeding Self-Efficacy Scale -Short form (BSES-SF) will be used to measure new mothers and father's breastfeeding self-efficacy. The mother breastfeeding self-efficacy was referred as a mother's confidence in her ability to breastfeed her infant, while the paternal breastfeeding self-efficacy was measured the father's confidence in his ability to support mothers' breastfeeding. The fathers version has been used previously. The BSES was originally developed by Dennis and Faux (1999) and has been translated into Chinese. It is a 14-item self-reported questionnaire with a 5-point scale that ranges from 1 to 5, with a total score ranging 5~70. A higher score represents a higher level of self-efficacy.The primary outcomes for this trial are commonly used breastfeeding indicators

SECONDARY OUTCOMES:
Exclusive breastfeeding rates | Change from Baseline Exclusive breastfeeding rates at 6 months.
  The primary outcomes for this trial are commonly used breastfeeding indicators
Anxiety symptoms | Change from Baseline Anxiety symptoms at 6 months.
  Anxiety symptoms of mother and her partner will be assessed using the Taiwanese version of the State Anxiety Inventory (SAI). The 20 item questionnaire contains a 4-point likert scale of 1 (not at all) to 4 (very much so), with an overall score ranging 20-80. A higher score indicates higher anxiety.
Depressive symptoms | Change from Baseline Depressive symptoms at 6 months.
  The Taiwanese version of the Edinburgh Postnatal Depression Scale (EPDS) will be used to assess depressive symptoms among new mother and father. EPDS has been used and tested in father participants with good validity. It is a 10-item self-reported questionnaire with a 4-point scale that ranges from 0 ("no") to 3 ("most of the time"), with a total score ranging 0~30. A higher score represents a higher level of depression. The suggested cutoff of 12/13 was used to detect probable cases of clinical depression, with a respective sensitivity and specificity of 83% and 89%.
Mindful awareness | Change from Baseline Mindful awareness at 6 months.
  The Five Facet Mindfulness Questionnaire at baseline, 1, 3 and 6 months The Taiwanese version of the Five Facet Mindfulness Questionnaire (FFMQ) will be adopted to assess new mothers' and partners mindfulness. The FFMQ has been translated into Chinese. It is a 39-item self-reported questionnaire with a 5-point scale that ranges from 1 (almost not) to 5 (almost always). A higher score represents a higher level of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Kuo, Doctoral, Principal Investigator — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei Medical University, Taiwan, R.O.C., Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseng JF, Chen SR, Au HK, Chipojola R, Lee GT, Lee PH, Shyu ML, Kuo SY. Effectiveness of an integrated breastfeeding education program to improve self-efficacy and exclusive breastfeeding rate: A single-blind, randomised controlled study. Int J Nurs Stud. 2020 Nov;111:103770. doi: 10.1016/j.ijnurstu.2020.103770. Epub 2020 Sep 3. PMID 32961461